CLINICAL TRIAL: NCT00551603
Title: Anaemia Correction in Haemodialyzed Patients - Comparative Analysis of Two Erythropoietin Stimulating Agents Schedules
Acronym: VAES
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistic reasons, financial contrastraints
Sponsor: Anemia Working Group Romania (Other)
Collaborators: Dr Carol Davila Teaching Hospital of Nephrology (Unknown); Romanian Renal Registry (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AWG_03_07; 1246/ANM
Record Dates: First submitted 2007-10-29; First posted 2007-10-31 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Bio-Equivalency of 2 Treatment Schedules in HD Patients
Keywords: epoetinum beta once-weekly; darbepoetinum once-fortnightly; anemia correction; hemoglobin stability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Group Epo will receive anaemia treatment according to the Romanian Best Practice Guidelines recommendation, with once-weekly SC epoetinum beta during the first phase, then will be switched to receive SC once-fortnightly darbepoetinum. Anaemia treatment schedule will continue according to the Romanian Best Practice Guidelines recommendations, with the same dose. A conversion factor of 1:200 will be used.
  Interventions: Drug: switch (epoetinum beta, darbepoetinum)
- 2 (Active Comparator): Subjects in the Darbepo Group will receive anaemia treatment according to the Romanian Best Practice Guidelines recommendation, with once-fortnightly or once-monthly darbepoetin SC administration, continuing their previous schedule and will continue their previous schedule of anaemia treatment during the second phase of the study
  Interventions: Drug: continuation (darbepoetinum)

INTERVENTIONS:
Drug: switch (epoetinum beta, darbepoetinum) — switching from epoetinum beta once weekly to once-fortnightly darbepoetinum
  Other Names: Group Epo
  Arms: 1
Drug: continuation (darbepoetinum) — continuation of the previous darbepoetinum administration schedule
  Other Names: Darbepo Group
  Arms: 2

SUMMARY:
Several recent reports support the efficacy of once every-other-week epoetinum administration in the maintenance phase of the anaemia treatment in predialysis, haemodialysis and in peritoneal dialysis CKD patients.

However, there are studies suggesting that in HD patients receiving SC short-acting ESA therapy, ESA efficacy decreases when the dosing is extended from thrice-weekly to once-weekly administration. When every-2-week administration of long-acting ESAs is extended to every 4 weeks, efficacy either remains stable or decreases incrementally. The GAIN trial (Gain effectiveness in Anemia treatment with NeoRecormon®) was designed to compare anemia management with epoetin beta, epoetin alpha or darbepoetin alpha in HD patients. An interim analysis of data from 1005 stable HD patients suggested that switching to epoetin beta from either epoetin alpha or darbepoetin alpha resulted in improved efficacy and a 20% dose reduction in SC epoetin beta.

The aim of the study is to compare two schedules of anaemia treatment in HD patients using two different erythropoietic stimulating agents (epoetinum beta vs darbepoetinum) with respect to the efficacy in anaemia correction and to the haemoglobin (Hb) level stability.

This is a multicenter (2 centers), prospective, open-label, parallel, controlled trial of therapy equivalence

DETAILED DESCRIPTION:
Currently available ESAs include epoetin alfa, epoetin beta, and darbepoetin. Epoetin alfa and beta have been designed to resemble closely the endogenous molecule and have similar pharmacokinetics. They are considered "short-acting" in comparison to darbepoetin, a second-generation molecule with a prolonged half-life, which is considered "long-acting." European and American Best Practice Guidelines (EBPG) recommend preferential subcutaneous (SC) twice- to thrice-weekly epoetin administration. There is a great deal of evidence that once-weekly SC administration of epoetin beta to be equally efficient and well tolerated in HD patients, even in those requiring high weekly epoetin doses. Several recent reports support the efficacy of once every-other-week epoetinum administration in the maintenance phase of the anaemia treatment in predialysis, haemodialysis and in peritoneal dialysis CKD patients.

However, there are studies suggesting that in HD patients receiving SC short-acting ESA therapy, ESA efficacy decreases when the dosing is extended from thrice-weekly to once-weekly administration. When every-2-week administration of long-acting ESAs is extended to every 4 weeks, efficacy either remains stable or decreases incrementally . The GAIN trial (Gain effectiveness in Anemia treatment with NeoRecormon®) was designed to compare anemia management with epoetin beta, epoetin alpha or darbepoetin alpha in HD patients. An interim analysis of data from 1005 stable HD patients suggested that switching to epoetin beta from either epoetin alpha or darbepoetin alpha resulted in improved efficacy and a 20% dose reduction in SC epoetin beta.

The aim of the study is to compare two schedules of anaemia treatment in HD patients using two different erythropoietic stimulating agents (epoetinum beta vs darbepoetinum) with respect to the efficacy in anaemia correction and to the haemoglobin (Hb) level stability.

The trial is designed according to the Guidelines for studies testing the equivalence of different treatment regimens , and will be conducted with the provisions of the Declaration of Helsinki and Tokio as amended in Venice (1983).

This is a multicenter (2 centers), prospective, open-label, parallel, controlled trial of therapy equivalence.

The total observation period is of 80 weeks:

* The baseline phase (pre-therapeutic intervention) - 12 weeks;
* The first study phase of therapeutical intervention - 48 weeks: each the two groups of patients will receive anaemia treatment according to the Romanian Best Practice Guidelines either with epoetinum beta or with darbepoetinum;
* The second study phase of therapeutical intervention - 24 weeks: the patients from the epoetinum beta group will be switched to darbepoetinum. The anaemia treatment will continue according to the Romanian Best Practice Guidelines, using the recommended conversion factor of 200 (Romanian Best Practice Guidelines, NKF-DOQI 2006, Revised EBPG).

  300 haemodialyzed patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* adult age (≥18 years)
* at least 6 months HD
* efficient HD (urea-equilibrated Kt/V >1.2, Daugirdas II equation)
* haemoglobin (Hb) levels above 10g/dL
* treatment with an ESA for at least 12 weeks prior to enrollment
* serum ferritin level 100-800 ng/mL
* transferrin saturation 20-50%.

Exclusion Criteria:

* hepatic diseases (as defined by abnormal ALT and AST levels) or association of psychical disorders or other disturbances making the enrollment unacceptable, as judged by the physician
* acute infection or HIV infection
* severe hyperparathyroidism (iPTH >800 ng/mL)
* active bleeding
* > 5% variation in dry body weight in the last 6 months
* previously diagnosed folic acid and/or vitamin B12 deficiency
* neoplastic diseases
* other known causes of anaemia
* known hypersensibility to one of the administered drugs
* epilepsy
* pregnancy or lactation
* anti-viral treatment during the month before the inclusion
* immunosuppressive treatment or use of other medication known to influence erythropoiesis during the month preceding the enrollment
* need for blood transfusions within 12 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
- hemoglobin level during the study and - monthly ESA dose per dry body weight during the study | 80 weeks of the study

SECONDARY OUTCOMES:
- percentage of patients maintaining target Hb without increase in ESA dose - difference between the average Hb during second study phase period versus the first one and versus baseline phase | during the study

CONTACTS AND LOCATIONS:
Overall Officials: Liliana Garneata, MD, PhD, Study Director — Anemia Working Group; Gabriel Mircescu, Professor, Study Chair — Anemia Working Group; Carmen Barbulescu, MD, Principal Investigator — "Dr Carol Davila" NephroCare Dialysis Centre; Alexandru Ciocalteu, Professor, Study Director — "IHS" Dialysis Centre "Sf Ioan Nou" Clinical Hospital; Daniela Ciortea, MD, PhD, Principal Investigator — IHS Dialysis Centre, "Sf Ioan Nou" Clinical Hospital
Locations (2):
- Romania (2):
  - "Dr Carol Davila" Fresenius NephroCare Dialysis Centre, Bucharest
  - IHS Dialysis Centre "Sf Ioan Nou" Clinical Hospital, Bucharest

REFERENCES:
- [Derived] Rath T, Mactier RA, Weinreich T, Scherhag AW; GAIN Investigators. Effectiveness and safety of recombinant human erythropoietin beta in maintaining common haemoglobin targets in routine clinical practice in Europe: the GAIN study. Curr Med Res Opin. 2009 Apr;25(4):961-70. doi: 10.1185/03007990902784459. PMID 19254204